CLINICAL TRIAL: NCT02845518
Title: EValuation of Cardiac Magnetic Resonance Imaging in Follow up assessmenT of Patients With Pulmonary Arterial Hypertension (EVITA)
Brief Title: Study of Cardiac MRI in the Follow up Assessment of Patients With PAH (EVITA)
Acronym: EVITA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, ARI CHAOUAT, Ari Chaouat (Associate Professor), Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PHRC-15-0210
Record Dates: First submitted 2016-06-21; First posted 2016-07-27 (Estimated); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary hypertension; right ventricular function; hemodynamics; prognosis
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- no arms (Experimental): All patients included will undergo a cardiac Magnetic Resonance Imaging (cMRI) at the baseline visit (V1), at 3- or 6-month follow up visit (V2 or V3), at 24-month follow up visit and in case of clinical worsening during the first 24-month of follow up.
  All patients will complete a questionnaire on the acceptability and tolerability of cMRI and right heart catheterization at V1, V2 or V3 and V9, right heart catheterization being performed as a routine test in pulmonary arterial hypertension.
  Depending on patient agreement, 22 ml of peripheral venous blood will be taken at visits V1, V2 or V3 and V9. On one of these 3 visits a blood sample of 5 ml will be taken from the pulmonary artery during the right cardiac catheterization.
  Interventions: Procedure: Cardiac magnetic resonance imaging (cMRI)

INTERVENTIONS:
Procedure: Cardiac magnetic resonance imaging (cMRI) — Right ventricular contouring and indexed aortic flow measurement from cMRI will be performed locally with the dedicated software used in clinical practice by the physicians of each centre. Cardiac index and RVEF will be derived from these measures. MRI interpretation will be performed blind with respect of clinical and RHC data.
  A self-administered questionnaire made up of 2 Likert scales will be given to all patients on visits V1, V2 or V3 and V9.
  To constitute a biobank for diagnosis and prognosis purposes blood samples will be taken at visits V1, V2 or V3 and V9.
  Other Names: Questionnaire; Blood samples

SUMMARY:
Pulmonary arterial hypertension (PAH) is characterized by a progressive increase in pulmonary vascular resistance leading to right ventricular failure and eventually to death. The therapeutic strategy has become complex and needs to perform recurring follow up evaluations including right heart catheterizations (RHC).

Cardiac magnetic resonance imaging (cMRI) has the advantage to accurately assess right ventricular volumes and important prognostic predictors such as cardiac index, stroke volume and right ventricular ejection fraction.

The main objective of EVITA is to assess the hemodynamic diagnosis performances at baseline and at follow up visits of cMRI in comparison with the results of the RHC (current guidelines) to detect an unfavorable hemodynamic status.

The primary endpoint is sensitivity and specificity of cMRI for the diagnosis of an unfavorable status defined by the current RHC criteria (with 95% confidence interval).

The secondary objectives are 1) to identify clinical and hemodynamic variables independently contributing to prognosis, 2) to describe complications due to cMRI and to RHC, 3) to compare acceptability and tolerability of cMRI over RHC for the patient, 4) to constitute biological collection of blood samples to determine diagnostic and prognostic PAH biomarkers, 5) To compare the measurements of indexed stroke volume performed by RHC and by cMRI, 6) To evaluate the prognostic value to predict an unfavourable hemodynamic status of cMRI variables (including indexed stroke volume) after taking into account NYHA functional class, 6-minute walk test distance and BNP or NT-proBNP after 4 months of PAH treatment and 7) To evaluate the prognostic value to predict the first occurrence of morbimortality events of cMRI variables (including indexed stroke volume) after taking into account NYHA functional class, 6-minute walk test distance and BNP or NT-proBNP after 4 months of PAH treatment.

PAH patients will be recruited in centers of the French network of severe pulmonary hypertension in a prospective cohort study.

180 subjects will be enrolled in the study: that size will give the study 90% power to find significant at the 5%-level.

If the primary endpoint were achieved, since first, strategies and procedures planed in this project are consistent with those currently used in routine and second, inclusion criteria are not limited to a sub-population of PAH patients, positive results could allow to broadly extend our findings.

Therefore, it will be possible to decrease the number of RHC, an invasive and cumbersome procedure without altering the prognosis. Moreover, all clinical procedures would be performed in outpatient clinics and thereby would reduce the cost to assess the severity of the disease. Current recommendations for evaluation of severity and follow-up being mainly derived from consensus of opinion of the experts, positive results will also improve the level evidence of severity assessment of PAH patients.

According to secondary objectives we expect to better predict morbimortality events with cMRI compared to RHC.

DETAILED DESCRIPTION:
Evaluation of cardiac magnetic resonance Imaging in follow up assessmenT of patients with pulmonary Arterial hypertension (EVITA) is a prospective cohort study of cMRI in PAH.

EVITA is a multicenter biomedical research study. All the investigation centers belong to the French network of severe pulmonary hypertension.

Pulmonary arterial hypertension (PAH) is characterized by a progressive increase in pulmonary vascular resistance leading to right ventricular (RV) failure and eventually to death. The therapeutic strategy has become complex and needs to perform recurring follow up evaluations including right heart catheterizations (RHC). Although, RHC performed in experience centers has low mortality and low morbidity, repeated invasive pulmonary hemodynamic measurements are burdensome and still presents some risk of complications. Once the diagnosis of PAH is established, follow up evaluation devoted to modifying specific therapy relies mainly on RV function parameters. Thus, echocardiography and cardiac magnetic resonance imaging (cMRI) meet many of the criteria of ideal monitoring tools.

Echocardiography is safe, inexpensive and widely available. However, this test has several limitations. Firstly, due to the complexity of the right ventricle chamber, the measurement of RV volumes is difficult. Secondly, criteria are numerous and for quantitative measurements different thresholds are applied without accepted definition. Thirdly, operator dependency could make it difficult to obtain reproducible images.

Cardiac MRI has the advantage to accurately assess RV volumes and important prognostic predictors such as cardiac index, stroke volume (SV) and right ventricular ejection fraction (RVEF).

It has been demonstrated that inter-observer and intra-observer variability for cMRI right ventricle measures in PAH patients were low. In addition, MRI-derived cardiac index, SV and RVEF significantly improved after few months of PAH specific therapy and had prognostic values regardless of changes of pulmonary vascular resistance in few trials of small size.

In a preliminary study performed in the CHRU-Nancy the investigators found in 21 subjects with PAH a significant correlation between cardiac output measured with cMRI and RHC (0.85, p<0.001). Furthermore, the agreement between the 2 methods was correct according to Bland-Altman plot.

The purpose of the present study is to investigate a strategy for assessing PAH severity. The investigators propose to replace a currently recommended method, i.e. RHC, by cMRI.

The researchers plan to use validated cardiac MRI measurements of RV volumes and cardiac output to demonstrate that cMRI can accurately assess the severity of the disease in a follow-up strategy.

The objectives of this project are to show that an assessment of the severity of the disease by a non-invasive pulmonary hemodynamic measurement using the cMRI is as effective as the RHC, and that it is reliable and safe.

The primary objective is to assess the performance of the cMRI (sensitivity and specificity) at baseline and during follow-up visits to detect an unfavorable hemodynamic state compared to the results of the RHC (current guidelines).

The secondary objectives are:

1. To assess the predictive value of the first morbi-mortality event in 2 different analyses derived, firstly from RHC criteria (cardiac index (CI)< 2.5 l/min/m² or a right atrial pressure > or = 8 mm Hg) and secondly from cMRI criteria (CI < 2.5 l/min/m² or RVEF < 35% or an absolute decrease of 10% of RVEF at a follow-up evaluation).
2. To assess the link between the first morbi-mortality event and New York Heart Association (NYHA) functional class, 6-minute walk distance, plasma level of B-type natriuretic peptide (BNP)/N-terminal(NT)-proBNP, and continuous hemodynamic variables from cMRI, RHC and echocardiography, data collected at baseline and after 3-6 months of follow-up in univariate analyses.
3. To assess the link between the first morbi-mortality event and the above factors, identifying clinical and hemodynamic variables independently contributing to prognosis in multivariate analyses. Using the results of this analysis the investigators plan to build a multiparameter prognostic score.
4. To quantify complications due to cMRI and to RHC.
5. To compare acceptability and tolerability of cMRI over RHC for the patient.
6. To create a biobank for diagnosis and prognosis purposes
7. To compare the measurements of indexed stroke volume performed by RHC and by cMRI.
8. To evaluate the prognostic value to predict an unfavourable hemodynamic status of cMRI variables (including indexed stroke volume) after taking into account NYHA functional class, 6-minute walk test distance and BNP or NT-proBNP after 4 months of PAH treatment.
9. To evaluate the prognostic value to predict the first occurrence of morbimortality events of cMRI variables (including indexed stroke volume) after taking into account NYHA functional class, 6-minute walk test distance and BNP or NT-proBNP after 4 months of PAH treatment.

This study is a prospective cohort study. PAH patients will be recruited in 20 centers of the French network of severe pulmonary hypertension.

A routine search for conditions known to cause pulmonary hypertension will be performed according to current guidelines. Therefore, all patients will undergo at baseline an echocardiography, an RHC and other routine tests.

A determination of NYHA functional class, BNP or NT-proBNP, 6-minute walk test and ECG 12 derivation should be performed at the earliest 2 days before the RHC during the screening period. As a reminder, RHC and cardiac MRI should be performed within 5 working days. Other examinations should be performed 12 months prior to the initial visit if the patient is prevalent, or 3 months prior to the initial visit if the patient is an incident patient.

If any specific PAH treatment is already in place (less than one year prior to the date of inclusion), it should be in stable dose for at least 1 month prior to the initial baseline visit.

This will be the screening period. Then all patients selected will sign the written informed consent of the main study, then the consent for the biobank if they accept them. The consent for the genetic study may be obtained at these visits or at a follow-up visit (no later than 24 months).

The collection of blood samples on one vein of the forearms for the biobank (and possibly for genetic analysis) will take place during this visit.

Subsequently, in the context of the study, a cMRI will be performed at the baseline visit (V1).

According to the current guidelines shortly after the baseline visit (V1) PAH-specific drug therapy will be initiated or associated to the treatment already in progress in incident cases or prevalent cases, respectively.

The follow-up period will be 24 months. A comprehensive severity evaluation will be performed after 3-6 months (V2 or V3) of the inclusion visit, after 24 months after the inclusion visit (V9) and in case of clinical worsening. According to current guidelines, these follow-up assessments will include NYHA functional class, 6-minute walk distance, plasma level of BNP/NT-proBNP and RHC. As part of one of the secondary objectives, 22 ml of venous blood will be collected during all RHC. During the visit 3-6 months (V2 or V3), 5 ml of blood from the pulmonary artery will be taken. Throughout the 24-month follow-up, patients will be seen on an outpatient basis every 3 or 6 months, depending on the practices of each center.

During the follow-up an echocardiography could be carried out at the discretion of the investigator at any visit in accordance with the current recommendations. According to the purpose of the present study, at all these visits a cMRI will also be performed.

All clinical procedures except cMRI and blood sample for the biobank, are those of standard care.

Morbidity and mortality will be collected prospectively until the last patient has completed his 24-month follow-up visit.

RHC will be performed according to currently recommended.

MRI data interpretation:

MRI protocol and post-processing guidelines will be sent prior to site initiation in order to apply the same method of cMRI in all centers. This will avoid important measurement error.

RV contouring and indexed aortic flow measurement will be performed locally with the dedicated software used in clinical practice by the physicians of each center. Cardiac index and RVEF will be derived from these measures. All cMRI images will be sent and stored at the CHRU Nancy. MRI interpretation will be performed blindly with respect of clinical and RHC data.

All adverse events will be collected during the follow up. The questionnaire assessing physical and psychological distress will be presented a few minutes after all RHC and all cMRI.

180 subjects will be enrolled in the study: that size will give the study 90% power to find significant at the 5%-level a sensitivity or specificity of:

* 90% with a lower 95% confidence limit of 75%,
* 60% with a lower 95% confidence limit of 40%.

General considerations:

Analysis of primary and secondary endpoints will be performed in the intention-to-treat and confirmatory analyses in the per-protocol populations. The 2-tailed significance level will set to p<0.05.

Analyses to respond to the main objective:

The aim of the trial is to assess the sensitivity and specificity cMRI regarding the diagnosis of unfavorable hemodynamic status determined from RCH measurements. Exact 95% confidence intervals of sensitivity and specificity will be computed.

Analyses to respond to secondary objectives:

Kaplan Meier life tables and curves will be produced as well as estimates of survival (morbi-mortality event) according to cMRI and RHC criteria given in the primary end point section.

Association between baseline factors and time to the first event of morbi-mortality will be assessed using Cox proportional hazard regression. Candidate factors will be identified among cMRI, RHC and echocardiography measurements along with NYHA functional class, 6-minute walk distance, plasma level of BNP/NT-proBNP and other potential baseline characteristics using univariable analysis. Factors found significant at the p<0.20 level will then be entered in a multivariable analysis with stepwise forward-backward selection. Only factors significant at the p<0.05 level will be kept in final multivariable model.

The same analyses will be repeated on data collected after 3-6 months of PAH specific treatment.

Complications of cMRI and RHC will be collected. The frequency of adverse events reported during the follow-up will be compared between groups using the Chi-Square test (or Fisher's exact test where requested).

Relative tolerability of cMRI and RHC will also be collected. The investigators will use the Kruskal-Wallis test to determine if the overall physical and psychological distress scores are different across the two groups.

Measurements of indexed stroke volume. Continuous variables (indexed stroke volume) will be compared by a paired t test.

Prognostic value. A multivariable model will be performed including all mentioned variables. The association of MRI variables with outcome will be assessed within the models. In addition, models with and without MRI variables will be compared with C-index and Net Reclassification Index (NRI) statistics to identify the added value of MRI variables.

If the primary endpoint were reached, positive results could allow to broadly extend our findings. Therefore, it will be possible to decrease the number of RHC, an invasive and cumbersome procedure without altering the prognosis. Positive results will also improve the level evidence of severity assessment of PAH patients.

According to the secondary objectives the investigators expect to better predict morbi-mortality events with cMRI compared to RHC. Thus, a composite score will be constructed including cMRI parameter and will be internally validated. Such a score can then be easily externally validated and widely used.

An ancillary study will be carried out in a few centers. This ancillary study is entitled "BI4P: BIomecanical Property of Pulmonary artery and Prognosis assessment in Pulmonary hypertension".

The main objective of BI4P is to assess the hemodynamic diagnosis performance of biomechanical parameters of the pulmonary artery at baseline and at follow up visits of 4D MRI to detect an unfavorable status in comparison with the results of the RHC.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age,
* Incident cases of PAH, or Prevalent cases of PAH diagnosed for less than 12 months when a re-evaluation is indicated including a right heart catheterization with the intention of modifying the specific-PAH treatment: from mono to dual therapy or from bi to triple therapy (if the 3rd treatment planned is parenteral epoprostenol, the centre must be able to perform an MRI under epoprostenol IV),
* Idiopathic, heritable PAH, or PAH associated with medication or toxic, or systemic scleroderma, or HIV infection or portal hypertension, or PAH associated with repaired (> 1 year) congenital systemic-to-pulmonary shunt.

Patients included in a biomedical trial to test a pharmaceutical treatment will be eligible provided that there is no incompatibility between the 2 studies.

Exclusion Criteria:

* Contraindication of cardiac MRI and impossibility to undergo MRI,
* Patients not in normal sinus rhythm at baseline,
* Patients with PH (pulmonary hypertension) due to left heart disease,
* Patients with PH due to lung diseases and/or hypoxemia,
* Chronic thromboembolic pulmonary hypertension,
* Comorbidities with a significant impact on the cardiovascular system such as valvulopathies, cardiomyopathy, severe hypertension despite appropriate treatment,
* Pregnancy,
* Patients under a measure of legal protection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-02-16 (Actual); Primary Completion 2024-05-16 (Estimated); Study Completion 2024-05-16 (Estimated)

PRIMARY OUTCOMES:
Performance of Cardiac Magnetic Resonance Imaging to detect an unfavorable hemodynamic state compared to the results of the Right Heart Catheterization | All visits will be pooled as one time point (unfavorable hemodynamic status from baseline to 24-month of follow up)
  Cardiac Magnetic Resonance Imaging CI < 2.5 l/min/m2 or a right ventricle ejection fraction (RVEF) < 35% or an absolute decrease of 10% of RVEF at a follow-up evaluation (for the second and third time-point) compared to cardiac index< 2.5 l/min/m2 or right atrial pressure > or = to 8 mm Hg measured with Right Heart Catheterization.

SECONDARY OUTCOMES:
Secondary objective 1: The predictive value of the first occurrence of morbimortality events in 2 different analyses derived from RHC criteria and from cMRI criteria. | From baseline to the end of the study. The end of the study is defined by the 24-month visit of the last patient included.
  The predictive value of the first occurrence of morbimortality events in 2 different analyses derived from RHC criteria and from cMRI criteria.
Secondary objective 2: The link between first morbimortality events occurrence and covariates, identifying variables independently contributing to prognosis in univariate analyses, to build a multiparameter prognostic score. | From baseline to the end of the study. The end of the study is defined by the 24-month visit of the last patient included.
  To assess the link between the first morbi-mortality event and the following factors (New York Heart Association (NYHA) functional class, 6-minute walk distance, plasma level of B-type natriuretic peptide (BNP)/N-terminal(NT)-proBNP, and continuous hemodynamic variables from cMRI, RHC and echocardiography), identifying clinical and hemodynamic variables independently contributing to prognosis in univariate analyses.
Secondary objective 3: The link between first morbimortality events occurrence and covariates, identifying variables independently contributing to prognosis in multivariate analyses, to build a multiparameter prognostic score. | From baseline visit to 24 month visit.
  To assess the link between the first morbi-mortality event and the following factors (New York Heart Association (NYHA) functional class, 6-minute walk distance, plasma level of B-type natriuretic peptide (BNP)/N-terminal(NT)-proBNP, and continuous hemodynamic variables from cMRI, RHC and echocardiography), identifying clinical and hemodynamic variables independently contributing to prognosis in multivariate analyses.
Secondary objective 4.a: Complications due to cMRI and to RHC | From baseline visit to 24 month visit.
  This will be mostly a descriptive analysis. The overall frequency of reported adverse events and severe adverse events will be compared between groups using the Chi-Square test (or Fisher's exact test where requested).
Secondary objective 4.b: Complications due to cMRI and to RHC | From baseline visit to 24 month visit.
  This will be mostly a descriptive analysis. The overall frequency of reported adverse events and severe adverse events will be compared between groups to account for the paired nature of the data, a McNemar test will be performed.
Secondary objective 5: The magnitude of better tolerability of cMRI over RHC for the patient | From baseline visit to 24 month visit.
  Physical and psychological distress due to cMRI and RHC will be measured with questionnaires.
  The comparison of the Likert-type scales of the questionnaires will be carried out using the Chi-Square test.
Secondary objective 6: Create a biobank for diagnosis and prognosis purposes | From baseline visit to 24 month visit.
  Blood samples to obtain DNA from circulating blood cells and plasma
Secondary objective 7: measurements of indexed stroke volume performed by RHC and by cMRI | From baseline visit to 24 month visit.
  Measurements of indexed stroke volume (in ml/m2) by RHC carried out at the same visit (baseline, 3-6 months, 24 months and visit in case of PAH worsening between 3-6 months and 24 months) than a cMRI exam.
Secondary objective 8: prognostic value to predict an unfavourable hemodynamic status of cMRI variables (including indexed stroke volume) after taking into account NYHA, 6-minute walk test distance and BNP or NT-proBNP after 4 months treatment | From baseline visit to 24 month visit.
  unfavourable status as defined for the primary objective.
Secondary objective 9: prognostic value to predict the first occurrence of morbimortality events of cMRI variables (including indexed stroke volume) after taking into account NYHA, 6-minute walk test distance and BNP or NT-proBNP after 4 months treatment | From baseline visit to 24 month visit.
  morbimortality as defined for the secondary objectives 1), 2) and 3).

CONTACTS AND LOCATIONS:
Overall Officials: CHAOUAT ARI, MD, PHD, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- Professor Ari CHAOUAT, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/18/NCT02845518/SAP_000.pdf